CLINICAL TRIAL: NCT02083757
Title: Fluid Responsiveness Predicted by Transcutaneous Partial Pressure of Oxygen in Critically Ill Patients
Brief Title: Fluid Responsiveness Predicted by PtcO2 in Critically Ill Patients
Acronym: PtcO2-FR
Status: Completed | Type: Observational
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Jingyuan,Xu, Zhongda Hospital, Southeast University, China
Other Study IDs: 2011ZDllKY03.0
Record Dates: First submitted 2014-03-07; First posted 2014-03-11 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Circulatory Failure
Keywords: Fluid responsiveness; Passive leg raising
MeSH Terms: conditions — Shock

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Resp: Fluid responsiveness is defined as a change of stroke volume stroke volume ≥ 10% after 250 ml rapid saline infusion in 10 minutes.
- Nonresp: Fluid responsiveness is defined as a change of stroke volume stroke volume < 10% after 250 ml rapid saline infusion in 10 minutes.

SUMMARY:
Our goal was to study the feasibility of predicting fluid responsiveness by transcutaneous partial pressure of oxygen (PtcO2) in the critically ill patients.

DETAILED DESCRIPTION:
The clinical determination of the intravascular volume can be extremely difficult in critically ill patients. Although hemodynamic maximization was proposed, this approach was associated with a risk of fluid overload and excessive inotropic support. Therefore, fluid optimization was seen as a significant step forward and has been shown to decrease complications. Significant effort has been devoted to defining and developing simple means for predicting fluid responsiveness, i.e. whether the patient will benefit from fluid administration. Passive leg raising (PLR), a bedside performed test, could be used to accurately predict fluid responsiveness in most conditions.

However, most parameters that provide information about fluid responsiveness during volume expansion and PLR are invasive and time-consuming. A completely noninvasive and atraumatic parameter to predict fluid responsiveness might be need urgently. Transcutaneous partial pressure of oxygen (PtcO2), a measure to detect tissue ischemia or inadequate perfusion, might reflect the change in cardiac output, thus predict fluid responsiveness. The purpose of this study was to study the feasibility of predicting fluid responsiveness by transcutaneous partial pressure of oxygen in the critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* clinical signs of inadequate tissue perfusion defined as systolic blood pressure < 90 mm Hg or a decrease > 40 mmHg in previously hypertensive patients or the need for vasopressive drugs (dopamine > 5 ug/kg/min or norepinephrine); urine output < 0.5 ml/kg/hr for 2 hrs; tachycardia; presence of skin mottling.

Exclusion Criteria:

* pregnancy, age of less than 18 years, contraindication to passive leg raising test, cardiac arrhythmias, cardiogenic pulmonary edema, the presence of abdominal compartment syndrome and refusal to participate in the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients for whom the attending physician decided to perform a fluid challenge or presence of at least one clinical sign of inadequate tissue perfusion in the absence of contraindication for fluid infusion for less than 24 hours were eligible to participate in the study.
Sampling Method: Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2011-09; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Cardiac Output | 30min
  Noninvasive bioreactance CO monitoring was obtained using the NICOM system (Cheetah Medical, Portland, OR) with four double-electrode stickers placed on the chest wall.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongda Hospital Southeast University, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Xu J, Peng X, Pan C, Cai S, Zhang X, Xue M, Yang Y, Qiu H. Fluid responsiveness predicted by transcutaneous partial pressure of oxygen in patients with circulatory failure: a prospective study. Ann Intensive Care. 2017 Dec;7(1):56. doi: 10.1186/s13613-017-0279-0. Epub 2017 May 23. PMID 28536944